CLINICAL TRIAL: NCT05529186
Title: Causes of Mortality in Kidney Transplant Recipients, a Paradigm Shift
Brief Title: Causes of Mortality in Kidney Transplant Recipients
Acronym: Paradigme
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8558
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Renal Disease
Keywords: renal disease; kidney transplant
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The causes of mortality in kidney transplant patients and the risk factors for mortality have been widely published. However, there is a high variability according to geographical areas and time. Recent studies suggest that the classical hierarchy of causes of mortality, i.e. the predominance of cardiovascular causes of death, could be overturned by the increase in infectious and cancer-related deaths. Investigators will try to highlight this paradigm shift and the related risk factors by studying two large French transplantation databases.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥18 years old) during transplantation
* Transplantation performed between 01/01/2008 and 31/12/2014
* Kidney transplant subject, double transplants kidney + pancreas, or kidney + islets of Langherans
* Subject previously transplanted other organs
* Subject not objecting, after being informed, to the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject having received a double transplant during the same operation: kidney + heart, kidney + liver, kidney + lungs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years old) with transplantation performed between 01/01/2008 and 31/12/2014
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Distribution of the causes of death of kidney transplant recipients presented in the form of percentage | Six months of starting dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Service Néphrologie-Dialyse-Transplantation - CHU de Strasbourg - France, Strasbourg, France